CLINICAL TRIAL: NCT01393379
Title: Effect of Endoscopic Lung Volume Reduction (ELVR) on Pulmonary Hypertension (PH) in Patients With Severe Emphysema and Pulmonary Hypertension
Brief Title: ELVR in PH Patients With Severe Emphysema
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Ekkehard Gruenig, Prof. Grünig / PD Dr. Eberhardt, Heidelberg University
Other Study IDs: S445/2009
Record Dates: First submitted 2011-07-12; First posted 2011-07-13 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: COPD; Pulmonary Emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pulmonary Emphysema

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate the effect of endoscopic valve implantation in patients with COPD and PH on hemodynamics, symptoms, exercise tolerance and quality of life in 10 patients in a prospective study. An improvement of objective parameters may also have a prognostic significance

DETAILED DESCRIPTION:
So far there is no treatment of COPD in addition to the established treatment of concomitant PH. Administration of PH-specific medication outside of clinical trials is not recommended in new guidelines for PH of the ERS/ESC. The influence of endobronchial valve implantation on the PH has not been studied in detail. The purpose of this study is to investigate the effect of endoscopic valve implantation in patients with COPD and PH on hemodynamics, symptoms, exercise tolerance and quality of life in 10 patients in a prospective study. An improvement of objective parameters may also have a prognostic significance

ELIGIBILITY:
Inclusion Criteria:

* signed patient consent form
* men and women >30 years
* Clinically indicated endoscopic lung volume reduction
* Pulmonary hypertension according to Group 3.1 of the Dana Point classification
* Severe pulmonary emphysema
* FEV1 <45%
* RV> 150%
* TLC> 100%
* Maximum of medical therapy according to GOLD
* heterogeneous emphysema
* Detected in the HR-CT
* Confirmation of the heterogeneity of emphysema by computer-assisted quantification (YACTA ®)
* stable COPD
* No exacerbation in the last 8 weeks
* Cortisone dose <20 mg prednisolone equivalent
* Non-or ex-smoker
* Nicotine abstinence> 4 months
* Actual CoHb <2.5%
* Diagnosis of pulmonary hypertension (PH), invasively diagnosed by right heart catheterization:
* Mean pulmonary arterial pressure (mPAP)> 25 mmHg
* Pulmonary capillary wedge pressure (PCWP) <15 mmHg
* Pulmonary vascular resistance (PVR)> 320 dyne * sec * cm-5

Exclusion Criteria:

* PH of Group 1, 2, 4, 5 of the Dana Point Classification
* Previous operations
* s/p Lung resection (lobectomy / pneumonectomy)
* s/p endoscopic lung volume resection
* significant bronchiectasis
* Sputum volume> 4 tablespoons / day
* Severe cardiac comorbidities:
* s/p myocardial infarction in the last 6 weeks
* Congestive heart failure
* Cardiomyopathy with highly impaired LVF
* Clopidogrel in long-term medication
* Respiratory insufficiency: PaCO2 mmHg at rest> 55
* current pregnancy

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe emphysema and PH, where ELVR is indicated
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-04; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Corvinus, MD, Principal Investigator — Center for pulmonary hypertension, Thoraxclinic Heidelberg
Locations (1):
- Center for pulmonary Hypertension, Thoraxclinic Heidelberg, Heidelberg, Germany